CLINICAL TRIAL: NCT03640195
Title: Acupoint Stimulation for Pain Reduction
Brief Title: Acupoint Stimulation for Pain Reduction and the Associated Benefits in Head and Neck Cancer Patients Receiving Concurrent Chemoradiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: yahe7693
Record Dates: First submitted 2018-07-11; First posted 2018-08-21 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-05

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Seeds

STUDY DESIGN:
Intervention Model Description: Intervention is divided into two parts: part of The Experimental group received Transcutaneous acupoint electrical stimulation 20 minutes/weeks, the acupoints are unilateral Hegu (LI4) and LU7; This study used Transcutaneous nerve electrical stimulation , 20 minutes each time, once a week for six consecutive weeks.
  The second part of The Experimental group received Auricular acupressure applied to four acupoints, including shenmen (TF2), mouth (IC6), subcortex (CW2), Occiput (AT3).A seeds embedding method with seeds attached to the four sides of the unilateral ear, using the thumb and forefinger to apply pressure, the participants will feel sour, each point is 1min, 5days/week, 3 times/day.
  Control group: without intervention
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Transcutaneous nerve electrical stimulation and Auricular acupressure.
  Interventions: Other: Device: Transcutaneous acupoint electrical stimulation and seeds for auricular acupressure
- Control group (No Intervention): without intervention

INTERVENTIONS:
Other: Device: Transcutaneous acupoint electrical stimulation and seeds for auricular acupressure — Experimental group received Acupoint stimulation, Transcutaneous acupoint electrical stimulation20 minutes/weeks, once a week for six consecutive weeks.
  The second part of The Experimental group received Auricular acupressure applied to four acupoints, including shenmen (TF2), mouth (IC6), subcortex (CW2), Occiput (AT3). each point is 1min, 5days/week, 3 times/day.
  Arms: Experimental group

SUMMARY:
This study was designed to investigate the effect of Acupoint stimulation on pain reduction, and fatigue, anxiety and depression and quality of life in Head neck cancer receiving Concurrent Chemoradiotherapy.

DETAILED DESCRIPTION:
Data were collected from 92 participants in northern Taiwan medical center Radiation Outpatient.They are randomly assigned to the experimental group (n=46) with Acupoint stimulation and control group(n=46). Outcomes were assessed according to the pain, Brief fatigue inventory, Hospital anxiety and depression scale, quality of life, five repeated measures was conducted.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of head and neck cancer with initial concurrent chemoradiotherapy
* Must be able to communicate clearly
* Must be above age 20

Exclusion Criteria:

* Previous radiotherapy
* History of arrhythmia or use of a pacemaker
* Local swelling or infection over the acupoint area

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-12-04 (Actual); Study Completion 2017-12-04 (Actual)

PRIMARY OUTCOMES:
Difference between the two groups from Baseline in Pain Scores on the Visual Analog Scale at 6 Weeks | from enrollment to end of treatment at 6 weeks
  Pain intensity was assessed using visual analogue scales (VAS) , which is a 10-cm continuous line to assess the subjective perception of pain in the case, with a score of 0 on the leftmost end of the line indicating "painless" and 10 points indicating The "most severe pain" and the reliability of pain assessment , and all participants received this linear tool measurement, recording a total of five

SECONDARY OUTCOMES:
Difference between the two groups from Baseline in fatigue on Brief Fatigue Inventory at 6 Weeks | from enrollment to end of treatment at 6 weeks
  Fatigue is using the friction fatigue inventory (BFI) ; it is a nitrate-item self-reported for measuring fatigue intensity and interference with functionality. Item 1-3 describes the fatigue strength, during The past 24 hour using a visual analogue scale (VAS) ranging from 0 (no fatigue) to 10 (very severely fatigued). Item 4-9 describes interferes with certain functions such as daily activity, including work, walking ability, normal work, Relations with others, and enjoyment in life. Each item was rated on a scale of 0 (does not interfere) to 10 (completely interferes). Its average score for each item indicates its severity of fatigue 1-3 points of helpful mild fatigue, 4 -6 is divided into moderate, 7-10 is divided into severe fatigue.
Difference between the two groups from Baseline in Anxiety and depression on Hospital Anxiety and depression scale | from enrollment to end of treatment at 6 weeks
  The Hospital Anxiety and depression scale (HADS) is composed of two seven-item subscales, one specifically targeting anxiety (HADS-A) and the other focusing on depression (HADS-D). The HADS is a 14-item measure divided into 2 subscales (anxiety and depression), HADS_A and HADS_D are scored separately, the topic arrangement is staggered, and the reverse problem is scored in reverse. The total score is between 0-21 points. Below 8 points means no anxiety and depression; 8 to 10 points may be anxiety and depression. And anxiety and depression of 10 points or more
Difference between the two groups from Baseline in quality of life European organization for research and treatment of cancer quality of life questionnaire head and neck 35(EORTC QLQ-H & N 35) | from enrollment to end of treatment at 6 weeks
  European organization for research and treatment of cancer quality of life questionnaire head and neck 35(EORTC QLQ-H & N 35) is a specific questionnaire developed by the European Organisation for Research and Treatment of Cancer for head and neck cancer. The module includes 35 questions Assessing symptoms and side effects of treatment, social function and body image/sexuality .This scale includes seven symptoms subscales that measure pain, swallowing, senses problems, speech problems, trouble with social eating, trouble with social Contact, and less sexuality, and also has 11 subscales related with teeth, opening mouth, dry mouth, sticky saliva, coughing, ill feeling, weight loss, weight gain, use of painkillers, nutritional supplements, and feeding tubes. Standardize the original scores, with scores ranging from 0 to 100, with higher scores representing more serious problems.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chou YH, Yeh ML, Huang TS, Hsu H. Acupoint stimulation improves pain and quality of life in head and neck cancer patients with chemoradiotherapy: A randomized controlled trial. Asia Pac J Oncol Nurs. 2021 Dec 25;9(1):61-68. doi: 10.1016/j.apjon.2021.11.002. eCollection 2022 Jan. PMID 35528798